CLINICAL TRIAL: NCT07250360
Title: Adjuvant Chemotherapy Confers Survival Benefit Only in High-Risk Pathologic Stage I Non-Squamous NSCLC: A Multicenter Prospective Cohort Study and Machine-Learning-Based Decision Tool
Brief Title: Adjuvant Chemotherapy for High-Risk Pathologic Stage I Non-Squamous NSCLC
Status: Completed | Type: Observational
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: No. 2024-SR-1028; No. 2024-SR-1028 (Other: Jiangsu Province Hospital)
Record Dates: First submitted 2025-09-28; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2024-02

CONDITIONS: Non-small Cell Lung Cancer Stage I
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 60 Months

GROUPS / COHORTS (2):
- Adjuvant chemotherapy
  Interventions: Drug: Adjuvant chemotheapy
- Postoperative Observation

INTERVENTIONS:
Drug: Adjuvant chemotheapy — apply adjuvant chemotheapy
  Groups: Adjuvant chemotherapy

SUMMARY:
Brief Summary The goal of this clinical trial is to evaluate the effect of postoperative adjuvant chemotherapy (ACT) in patients with stage I non-squamous non-small cell lung cancer (NSCLC) after curative resection.

The main questions it aims to answer are:

Does ACT improve recurrence-free survival (RFS) compared with observation alone?

Does ACT provide disease-free survival (DFS) benefit in this patient population?

Researchers will compare the adjuvant chemotherapy group with the observation group to see if chemotherapy reduces the risk of recurrence and improves survival outcomes.

Participants will:

Receive standard platinum-based adjuvant chemotherapy after surgery or undergo regular postoperative surveillance according to institutional guidelines.

Be followed at scheduled intervals with clinical assessments and imaging to monitor for recurrence and survival outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must have histologically confirmed non-squamous NSCLC
2. Patients must be ≥18 years of age at the time of diagnosis
3. Pathological stage I disease (T1-2N0M0) according to the AJCC 8th edition (specify if applicable)
4. Patients must have undergone complete surgical resection (R0) with systematic lymph node dissection
5. Surgery performed between January 1, 2015 and December 31, 2019

Exclusion Criteria:

1. Prior history of malignant tumors or presence of synchronous other primary malignancy
2. Multiple primary lung cancers diagnosed at baseline
3. Receipt of any neoadjuvant chemotherapy, radiotherapy, or targeted therapy
4. Perioperative death occurring within 30 days after surgery
5. Incomplete or missing clinical or pathological information
6. Loss to follow-up before the first scheduled surveillance assessment

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: patients with non-squamous NSCLC from four participating hospitals
Sampling Method: Non-Probability Sample
Enrollment: 2072 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2019-12-31 (Actual); Study Completion 2025-06-01 (Actual)

PRIMARY OUTCOMES:
5-year Disease-Free Survival (DFS), defined as time from surgery to recurrence or death, estimated by Kaplan-Meier method. | Up to 5 years after surgery
  DFS is defined as the time from surgery to the first documented recurrence or death from any cause, whichever occurs first. Patients without an event will be censored at the last follow-up. Data will be summarized using Kaplan-Meier survival analysis, with median DFS and 95% confidence intervals.

SECONDARY OUTCOMES:
5-year Recurrence-Free Survival (RFS), defined as time from surgery to the first recurrence or death from any cause, estimated by Kaplan-Meier method | Up to 5 years after surgery.
  RFS is defined as the time from surgery to the date of first documented tumor recurrence (local, regional, or distant) or death from any cause, whichever occurs first. Patients who are alive and recurrence-free will be censored at the date of last follow-up. Data will be analyzed using Kaplan-Meier survival estimates, with median RFS and 95% confidence intervals reported.